CLINICAL TRIAL: NCT04809116
Title: Open-label Pimavanserin 34mg at Bedtime for 6 Weeks for Insomnia in Veterans With Post-traumatic Stress Disorder: Proof of Concept Study
Brief Title: Pimavanserin for Insomnia in Veterans With Posttraumatic Stress Disorder: Proof of Concept
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Received alternative sources of funding.
Sponsor: Baylor College of Medicine (Other)
Collaborators: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Principal Investigator, Melissa Jones, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-48699
Record Dates: First submitted 2021-03-15; First posted 2021-03-22 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Insomnia Chronic; Posttraumatic Stress Disorder
Keywords: insomnia; posttraumatic stress disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Stress Disorders, Post-Traumatic | interventions — pimavanserin

STUDY DESIGN:
Intervention Model Description: open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- open-label pimavanserin 34mg at bedtime for 6 weeks (Experimental): Subjects enrolled into treatment with open-label, fixed-dose pimavanserin 34mg at bedtime for 6 weeks
  Interventions: Drug: Pimavanserin

INTERVENTIONS:
Drug: Pimavanserin — open-label, fixed-dose pimavanserin 34mg at bedtime for 6 weeks
  Other Names: Nuplazid

SUMMARY:
This is a proof-of-concept, open-label trial of pimavanserin 34mg at bedtime for 6 weeks in Veterans with insomnia and Posttraumatic Stress Disorder.

DETAILED DESCRIPTION:
More treatments are needed to target insomnia in Veterans with Posttraumatic Stress Disorder. There is evidence to suggest that pimavanserin, a medication approved by the Food and Drug Administration for the treatment of psychosis in Parkinson's disease, may improve deep sleep and insomnia. This proof-of-concept study preliminarily assesses the feasibility of open-label, fixed-dose pimavanserin 34mg at bedtime for 6 weeks for the treatment of chronic insomnia in Veterans with Posttraumatic Stress Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Veterans, aged 18-64
* Determined to meet criteria for current posttraumatic stress disorder, as per the Clinician Administered PTSD Scale for the DSM-5 (CAPS-5) and a total score of ≥33 on the PTSD Checklist (PCL-5)
* Meets DSM-5 standards of chronic insomnia disorder, as follows: a. Complains of dissatisfaction with nighttime sleep in the form of difficulty falling asleep (subjective sleep onset latency ≥30 minutes), difficulty staying asleep (subjective time awake after sleep onset ≥30 minutes), and/or awakening earlier in the morning (≥30 minutes before scheduled wake time and before a total sleep time of 6.5 hours) than desired. b. Insomnia frequency of ≥3 times per week c. The duration of the insomnia complaint is ≥3 months d. Associated with complaint of daytime impairment
* Insomnia Severity Index total score ≥15 (moderate insomnia)
* Willing and able to comply with all aspects of the protocol
* Willing to not start a concurrent behavioral or other treatment program for insomnia, PTSD, or other psychiatric disorders during the participation in the study
* If female subjects nor their partners are surgically sterile, and if they are not post- menopausal (absence of menses for at least 12 months), female subjects are considered to be of child-bearing potential. It is required that women of child-bearing potential who are sexually active agree to either refrain from sexual activity or use a two methods of contraception for the duration of the study (i.e., beginning 30 days prior to drug initiation and extending to 30 days after the last dose of study drug). The two methods should include: 1) A barrier method (e.g., condom with spermicidal gel, diaphragm with spermicide, intrauterine devices, cervical cap), and 2) One other method, including hormonal contraceptives (e.g., oral contraceptives, injectable contraceptives, contraceptive implant) or another barrier method.

Exclusion Criteria:

* Current or a history of a primary psychotic disorder (i.e., schizophrenia, schizoaffective or bipolar disorder)
* Active suicidal or homicidal ideation requiring crisis intervention
* Current moderate or severe alcohol or marijuana/cannabis use disorder, or other illicit use disorder of any severity
* A history of moderate or severe traumatic brain injury or other neurological illness (i.e., stroke, epilepsy, multiple sclerosis)
* Caffeine use that is deemed excessive and is contributing to the insomnia per the opinion of the investigators (i.e. caffeinated beverages consumed after 18:00 3 times/week or more and/or that correlates with the timing of the insomnia complaints)
* Tobacco use before bedtime that is contributing to the insomnia per the opinion of the investigators or that would interfere with completing an overnight polysomnogram
* Previous diagnosis of periodic limb movement disorder, restless legs syndrome, circadian rhythm sleep disorder, narcolepsy, RBD, or other sleep disorders (except obstructive sleep apnea) that may confound, per the opinion of the investigators, the assessment of insomnia
* Previous diagnosis of moderate to severe obstructive sleep apnea (defined as an AHI equal to or greater than 15)
* Participants deemed to be at high risk of moderate to severe obstructive sleep apnea per the Snoring, Tiredness, Observed apnea, high blood Pressure, Body mass index, Age, Neck circumference, and male Gender questionnaire (STOP-BANG). Subjects with a STOP-BANG score of 5 or greater, or STOP score of 2 or greater plus (body mass index greater than 35 kg/m2 or male or neck circumference greater than 40 cm), are considered to be high-risk and will be referred to clinical treatment
* Participants identified as having moderate to severe obstructive sleep apnea during the screening polysomnogram. These participants will be referred to clinical treatment
* Periodic limb movement arousal index 15 or greater or other sleep disorders captured during the screening polysomnogram that may confound, per the opinion of the investigators, the assessment and treatment of insomnia
* A prolonged QT interval, corrected for heart rate (QTc), at the screening electrocardiogram. A prolonged QTc is defined as 470 milliseconds for males and 480 milliseconds for females
* Engagement in an evidence-based psychotherapy within 1-week prior to enrollment that in the opinion of the investigators, may confound the assessment of insomnia (ex. CBT for insomnia)
* Current evidence of clinically significant cardiac, respiratory, gastrointestinal, renal, neurological, hepatic, and/or chronic pain that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments
* Females who are breastfeeding or pregnant at screening; 16. Females of childbearing potential who are not practicing acceptable pregnancy prevention methods (NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal or have been sterilized surgically)
* Patients with cardiac conditions that in the opinion of the investigators may increase the risk of torsades de pointes and/or sudden death (ex. symptomatic bradycardia, congenital prolongation of the QT interval)
* Current use of a prohibited medications: Hypnotic or sedating medications taken at bedtime for insomnia; antipsychotics and antidepressants with known 5HT2A antagonist activity; medications that increase or decrease the metabolism of pimavanserin; medications that increase the risk of QTc prolongation

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates | 7 months
  The number of subjects enrolled into treatment per month; goal of 20 total
Retention rates | 12 months
  The number of subjects completing treatment; goal of 16 (80%)

SECONDARY OUTCOMES:
Mean change in duration of stage N3 sleep pre- and post-treatment | 6 weeks
  The mean change in duration of stage N3 sleep from baseline polysomnogram to week-6 polysomnogram
Discontinuation rates due to adverse effects | 12 months
  The number of subjects who discontinue the protocol due to adverse effects
Completion rates of key outcome measures | 12 months
  The percentage of participants who complete subject and objective measures of insomnia, including sleep diaries, actigraphy, and attended polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Melissa B Jones, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No